CLINICAL TRIAL: NCT02216487
Title: Phase II Single Arm Trial of FOLF(HA)Iri Plus Cetuximab in Irinotecan-naïve Second Line Patients With KRAS Wild Type Metastatic Colorectal Cancer
Brief Title: Trial of FOLF(HA)Iri With Cetuximab in mCRC
Acronym: Chime
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Western General Hospital, Australia (Other)
Collaborators: Alchemia Oncology (Industry); Merck Serono International SA (Industry)
Responsible Party: Principal Investigator, Peter Gibbs, Associate Professor, Western Hospital, Australia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACO-004
Record Dates: First submitted 2014-08-12; First posted 2014-08-15 (Estimated); Last update posted 2014-08-29 (Estimated); Status verified 2014-08

CONDITIONS: Metastatic Colorectal Cancer
Keywords: mCRC; colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- HA-Irinotecan (Experimental): HA-Irinotecan is administered as part of FOLFIRI/cetuximab treatment in place of irinotecan.
  Interventions: Drug: HA-Irinotecan

INTERVENTIONS:
Drug: HA-Irinotecan — HA-Irinotecan is administered as part of FOLFIRI/cetuximab treatment in place of irinotecan for treatment of mCRC.

SUMMARY:
As an approach to improve efficacy and provide clinical benefit to cancer patients undergoing chemotherapeutic treatment regimens, Alchemia Oncology has developed a novel means for delivering anti-cancer agents to tumours. The drug delivery platform is based on the use of hyaluronic acid (HA), a novel excipient, in which, formulation with HA results in optimisation of cytotoxic drug uptake and retention within solid tumours. In the specific example of HA-Irinotecan, this new formulation of irinotecan has demonstrated enhanced efficacy in both nonclinical and early clinical studies.

The current study is an investigation into the use of HA-Irinotecan in a Phase II single arm trial of FOLF(HA)iri plus cetuximab in irinotecan-naïve second line patients with KRAS wild type metastatic colorectal cancer. The study objectives are to confirm the safety and efficacy of FOLF(HA)iri plus cetuximab as second-line therapy in irinotecan-naïve metastatic colorectal cancer patients.

It is expected that the study recruit approximately 40-50 patients in 1 year with subsequent treatment and follow up; thus the trial will run for approximately 2-3 years.

ELIGIBILITY:
Inclusion criteria

* Tumour is KRAS wild type
* mCRC with disease progression after first-line chemotherapy (adjuvant chemotherapy is considered first line chemotherapy if metastatic progression occurs within 6 months of the end of the adjuvant chemotherapy).
* Irinotecan naïve
* Prior use of bevacizumab in the 1st line setting is permitted.
* ECOG 0 or 1
* Measurable disease
* Histological proof of colorectal adenocarcinoma
* 18+ years of age
* Adequately recovered from and at least 4 weeks after recent major surgery or chemotherapy
* At least 4 weeks after treatment with a biologic monotherapy from last dose to enrolment.
* Hematology done within 14 days prior to enrolment :

  * Absolute Neutrophil count (ANC) greater than 1.5 x 109/L
  * Platelets greater than 100 x 109/L
  * Hemoglobin greater than or equal to 100g/L
* Chemistry done within 14 days prior to enrolment:

  * AST greater than or equal to 2.5 X ULN (greater than 5 X ULN if elevation thought to be related to hepatic metastatic disease),
  * Alkaline phosphatase greater than 5 x ULN,
  * Serum creatinine greater than 1.5 x ULN,
  * Total bilirubin greater than 34.2 µmol/L,
  * Negative serum or urine pregnancy test if a WOCBP.

Exclusion criteria

* KRAS mutant.
* Prior irinotecan
* Prior anti-EGFR
* History of other malignancies, except adequately treated non-melanoma skin cancer, curatively treated in-situ cancer of the cervix, or other solid tumours curatively treated with no evidence of disease for greater than 5 years.
* Locally advanced or recurrent disease only
* Unsuitability for irinotecan
* Abdominal or pelvic radiation therapy (including treatment with SIR-Spheres/Sirtex) within the last 12 months.
* Women who are pregnant or breastfeeding.
* Significant cardiac disease
* Untreated or symptomatic brain or central nervous system (CNS) metastases
* Presence of pleural effusion or ascites requiring therapeutic thoracocentesis or paracentesis.
* Current partial or complete bowel obstruction.
* Concomitant active infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2014-06; Primary Completion 2016-06 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Safety | 2 years
  To assess FOLF(HA)iri plus cetuximab with respect to:
  Patient safety, including incidence of severe (Grade 3/4) toxicity according to the National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI CTCAE version 4.03).

CONTACTS AND LOCATIONS:
Overall Officials: Peter Gibbs, MD, Principal Investigator — Western General Hospital
Locations (3):
- Australia (3):
  - Liverpool Hospital, Sydney, New South Wales
  - Southern Medical Day Care Centre, Wollongong, New South Wales
  - Western General Hospital, Melbourne, Victoria